CLINICAL TRIAL: NCT02188615
Title: A Single Institution Prospective Randomized Controlled Clinical Trial of Neo-adjuvant Chemoradiotherapy Followed by Mckeown Minimally Invasive Esophagectomy (MIE) Versus Mckeown MIE for Locally Advanced Squamous Cell Esophageal Carcinoma
Brief Title: Study of Neo-adjuvant Chemoradiotherapy Followed by Minimally Invasive Esophagectomy for Squamous Cell Esophageal Cancer
Acronym: NACRFMIE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengchu Zhu (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other)
Responsible Party: Sponsor-Investigator, Chengchu Zhu, Division Director, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BZhang; 2011C13039-2 (Other Grant/Funding Number: Zhejiang Provincial Science and Technology Major Projects)
Record Dates: First submitted 2014-06-28; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Squamous Cell Esophageal Carcinoma
Keywords: Squamous Cell Esophageal Carcinoma; minimally invasive esophagectomy; laparoscopy; thoracoscopy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Vinorelbine; Thoracoscopy; Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- experimental group (Experimental): Neo-adjuvant Chemoradiotherapy followed by Mckeown MIE
  Interventions: Procedure: Neo-adjuvant Chemoradiotherapy followed by Mckeown MIE
- Radical Chemoradiotherapy (Active Comparator): only Radical Chemoradiotherapy
  Interventions: Drug: Cisplatin
- Mckeown MIE (Active Comparator): only Mckeown MIE
  Interventions: Device: Mckeown MIE

INTERVENTIONS:
Procedure: Neo-adjuvant Chemoradiotherapy followed by Mckeown MIE — Neo-adjuvant Chemoradiotherapy followed by Mckeown MIE
  Arms: experimental group
Drug: Cisplatin — only Radical Chemoradiotherapy
  Other Names: vinorelbine
  Arms: Radical Chemoradiotherapy
Device: Mckeown MIE — only Mckeown MIE using thoracoscopy and laparoscopy
  Other Names: Thoracoscopy; Laparoscopy
  Arms: Mckeown MIE

SUMMARY:
The primary objective is to compare neo-adjuvant chemoradiotherapy followed by Mckeown Minimally Invasive Esophagectomy (MIE) Versus Mckeown MIE, pure radical chemoradiotherapy in terms of the overall survival time (OS) in patients with Stage IIB or III squamous cell esophageal carcinoma.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most difficult malignancies to cure. Surgical resection remains the primary treatment for localized esophageal cancer. It increases the chances of cure and alleviates the symptoms of dysphagia compared with nonoperative methods. Advances in surgical techniques and equipments have made minimally invasive esophagectomy (MIE) more popular and wider application since 1990s. During the past two decades, MIE has progressively been accepted as an alternative treatment for esophageal cancer around the world. The prognosis has some improvement on account of these significant advances in surgical techniques and perioperative management, But the prognosis of patients with locally advanced esophageal cancer remains rather poor. As a result of surgery alone, the 5-year survival rate of about 25% has not changed significantly in several decades.

Preoperative chemoradiotherapy followed by surgery seems to hopefully improve the survival of EC. Nevertheless, the results of different studies were inconsistent. Recently, the CROSS trial has demonstrated that preoperative chemoradiotherapy can significantly increased the overall survival of patients with EC compared with surgery alone. It should be noticed that only 84 cases(23%) of ESCC were enrolled in this trial with potential minimal follow-up of 2 years, which may be not perfect to evaluate the effect of this combined therapy for this tumor type.

Based on our preliminary study, we have demonstrated the validity and safety of vinorelbine and cisplatin-based neoadjuvant chemoradiotherapy. Then we are to carry out a clinical trial to investigate the effect of this multidisciplinary therapy, by comparing neo-adjuvant chemoradiotherapy followed by Mckeown MIE versus Mckeown MIE, pure radical chemoradiotherapy in terms of the overall survival time (OS) in patients with Stage IIB or III squamous cell esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage IIB or III, which is potentially resectable.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival.
4. Age ranges from 18 to 70 years.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. Karnofsky performance status (KPS) of 90 or more.
7. Signed informed consent document on file.

Exclusion Criteria:

1. Patients are diagnosed or suspected to be allergic to cisplatin or vinorelbine.
2. Patients with concomitant hemorrhagic disease.
3. Pregnant or breast feeding.
4. Inability to use gastric conduit after esophagectomy because of a prior surgery.
5. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more.
6. Have a prior malignancy other than esophageal carcinoma, carcinoma in situ of the cervix, nonmelanoma skin cancer or cured early stage of prostate cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 1 years
Disease free survival | 5years
Overall survival rate | 3years
Overall survival rate | 5years

SECONDARY OUTCOMES:
the opportunity of MIE after neo-adjuvant chemoradiotherapy | 4 weeks after completion of radiotherapy
  Criteria:Response Evaluation Criteria in Solid Tumors，RECIST
Side effects of neo-adjuvant chemoradiotherapy | 2 weeks after completion of radiotherapy
  Evaluate the toxicities of neo-adjuvant chemoradiotherapy,according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 3.0
Duration of surgery | Intraoperative
  The time between the start of surgery until the end of surgery
Quantity of bleeding | Intraoperative
  The amount of bleeding during surgery
number of lymph nodes retrieved | Intraoperative
  The total number of lymph nodes obtained including cervix area, mediastinum area , abdominal area
Days of postoperative stay | The duration of hospital stay after surgery, an expected average of 12 days
  Participants will be followed for the duration of hospital stay after surgery, an expected average of 12 days
Rate of Operative Complication | 30 days after surgery
Mortality of perioperation | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cheng chu Zhu, professor, Study Chair — Taizhou Hospital; Bao fu Chen, professor, Study Director — Taizhou Hospital
Locations (1):
- Thaizhou Hospital, Linhai, Zhejiang, China